CLINICAL TRIAL: NCT04877262
Title: Effects of Time-restricted Eating on Nutrient Absorption in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Claire E. Berryman, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001564
Record Dates: First submitted 2021-03-14; First posted 2021-05-07 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Digestibility
Keywords: stool energy loss; digestibility; intestinal absorption; overweight; microbiome; metabolomics; energy balance
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: The study is a randomized, crossover, controlled feeding study design consisting of two 9-d weight maintenance diet periods separated by at least 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early time-restricted eating (eTRE) (Experimental): Participants will be provided a weight-maintenance diet for 9 consecutive days and will consume all meals and snacks in a 6-h window in the morning hours (e.g., 8:00 AM - 2:00 PM)
  Interventions: Other: weight maintenance diet (WMD)
- control eating schedule (CON) (Experimental): Participants will be provided a weight-maintenance diet for 9 consecutive days and will consume all meals and snacks in a 12-h window in the morning hours (e.g., 8:00 AM - 8:00 PM)
  Interventions: Other: weight maintenance diet (WMD)

INTERVENTIONS:
Other: weight maintenance diet (WMD) — A diet meeting the participant's weight maintenance energy needs will be provided.

SUMMARY:
This 2-period, crossover, controlled-feeding trial will investigate the effects of early time-restricted eating (8am-2pm), compared to a control eating timeframe (8am-8pm), on energy and macronutrient digestibility, the thermic effect of food (TEF), postprandial blood metabolites, 24 h glucose concentrations, glycemic variability, intestinal hydrogen gas production, gastrointestinal transit time, and microbiome composition. This study will also seek to determine factors that may predict intestinal absorption efficiency (i.e., digestibility) including the microbial composition of stool, fasting and postprandial metabolomics, gastrointestinal transit time, thermic effect of food, 24 h glucose concentrations and variability, and hydrogen gas production.

DETAILED DESCRIPTION:
The obesity epidemic is well documented, and despite a complex etiology influenced by genetic, physiological, psychological, social, behavioral, and environmental factors, obesity seems to be the result of energy imbalance, where energy intake exceeds energy expenditure, regardless of the internal and external influences. Studies aiming to quantify and manipulate modulators of energy balance, including gastrointestinal (GI) energy absorption rates (i.e., digestibility), are crucial for reducing the incidence of overweight and obesity and improving overall human health. Despite considerable interindividual variability in the amount of ingested energy that is absorbed (~87-98% of ingested energy) by the gastrointestinal tract, generalized equations are used to calculate individual energy intake requirements, and the factors that contribute to such variability, including meal-timing, are largely unknown.

The proposed study seeks to determine the effects of restricting the eating window to 6-h (early time-restricted eating) as compared to a control eating window of 12 h on energy and macronutrient digestibility, thermic effect of food (TEF), postprandial blood metabolites (triglyceride, insulin, glucose, fructose, galactose, inositol, and sorbitol), 24 h glucose concentrations and glycemic variability, intestinal hydrogen gas production, microbiome composition, and gastrointestinal transit time in response to a controlled, energy balanced diet. In addition, this project will determine whether energy digestibility can be predicted from biological and physiological factors such as gut microbiota composition, gastrointestinal transit time, 24-h glucose concentrations, and postabsorptive and postprandial metabolomic profiles.

Participants will be randomized to early TRE (6-h feeding window, 8am-2pm) or a control eating schedule (12-h feeding window, 8am-8pm) and consume a controlled, energy balance diet (breakfast, lunch, dinner, snacks, and beverages) for 9 consecutive days before crossing over to the other intervention after at least a 3-wk washout for females (to control for hormonal fluctuations) and at least a 2-wk washout for males. Participants will collect stool and urine during each feeding phase. Gross energy content (heat combustion by bomb calorimetry) of the diet, stool, and urine samples will be used to calculate energy digestibility (diet gross energy - stool gross energy) and metabolizable energy. Factors that may mediate and/or predict energy digestibility efficiency, including gastrointestinal microbial composition, transit time, and gas production, fasting and postprandial metabolites, continuous glucose concentrations, and thermogenesis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years old
* Normal weight or overweight (18.5 to 29.9 kg/m2)
* Not taking any probiotics for 4 weeks prior to and throughout the entire study
* Willing to refrain from smoking, vaping, chewing tobacco, and dietary supplement use throughout the study
* Willing to consume a controlled diet for 9 consecutive days on 2 different occasions (18 days total) and collect all urine and fecal output for 3-5 days during each occasion
* Pass the blue dye gastrointestinal tracer (given at screening) within 72 hours of administration

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, prior bariatric surgery, malabsorption, or any condition that interferes with metabolism (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Suspected or known strictures, fistulas, or physiological/mechanical gastrointestinal obstruction
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Women who are pregnant, lactating, planning to become pregnant, or who have an irregular menstrual cycle in the past 6 months
* Weight fluctuations ± 5% of body weight in the last 6 months
* Allergies or intolerance to foods included in the controlled diet
* Any use of antibiotics, except topical antibiotics, within 3 months of study participation
* Colonoscopy within 3 months of study participation
* Use of laxatives, stool softeners, or anti-diarrheal medications more than once a week within 4-weeks of study enrollment

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Energy digestibility | Days 4-9
  Calculated as gross energy of the diet (kcals) - gross energy excreted in stool (kcals)

SECONDARY OUTCOMES:
Fat digestibility | Days 4-9
  Calculated as fat content of the diet - fat content excreted in stool
Carbohydrate digestibility | Days 4-9
  Calculated as carbohydrate content of the diet - carbohydrate content excreted in stool
Protein digestibility | Days 4-9
  Calculated as protein content of the diet - protein content excreted in stool
Metabolizable energy | Days 4-9
  Calculated as gross energy of the diet (kcals) - gross energy excreted in urine and stool (kcals)
Metabolizable protein | Days 4-9
  Calculated as protein content of the diet - protein excreted in urine and stool
Postabsorptive and postprandial plasma metabolites | Day 6
  Plasma metabolites will be measured using gas chromatography coupled with mass spectrometry in the postabsorptive state and following a standardized meal (1 hour, 2 hours, 3 hours, and 4 hours after meal intake).
Gut microbiome | Day 6
  Microbiota composition and diversity will be determined using 16S rRNA gene sequencing.
Gastrointestinal transit time | Day 6
  A gas-sensing capsule will be ingested to measure transit time in the gastrointestinal tract.
Gastrointestinal gas production | Day 6
  A gas-sensing capsule will be ingested to measure hydrogen, carbon dioxide, and oxygen production in the gastrointestinal tract.
Gastrointestinal temperature | Day 6
  A gas-sensing capsule will be ingested to measure temperature in the gastrointestinal tract.
24-h glucose concentrations | Days 1-8
  A continuous glucose monitor will be used to collect and assess 24-h glucose concentrations.
24-h glucose variability | Days 1-8
  A continuous glucose monitor will be used to collect and assess 24-h glucose variability.
Thermic effect of food | Day 6
  Indirect calorimetry measures will be collected in the resting state and for 4 hours (15-30, 45-60, 75-90, 105-120, 165-180, and 225-240 minutes) following the consumption of a standardized meal.

CONTACTS AND LOCATIONS:
Overall Officials: Claire E Berryman, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson MA, Cheung SN, La Frano MR, Nagpal R, Berryman CE. Intestinal Energy Absorption Is Associated with Glycemic Variability in Young, Healthy Adults. J Nutr. 2025 Jul;155(7):2205-2214. doi: 10.1016/j.tjnut.2025.05.018. Epub 2025 May 23. PMID 40414300
- [Derived] Dawson MA, Cheung SN, La Frano MR, Nagpal R, Berryman CE. Early time-restricted eating improves markers of cardiometabolic health but has no impact on intestinal nutrient absorption in healthy adults. Cell Rep Med. 2024 Jan 16;5(1):101363. doi: 10.1016/j.xcrm.2023.101363. PMID 38232698